CLINICAL TRIAL: NCT02942121
Title: Application-based Perioperative Management of the Radical Cystectomy Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: University of Kansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003585
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Bladder Cancer
Keywords: surgery education; radical cystectomy; cystectomy; muscle-invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LST App (Experimental): Participants will use the LifeScience Technologies application (LST app) before surgery, and post surgery. Participants will use the app as an educational tool to learn more about their surgery. Participants will also answer questions about themselves in the app.
  Interventions: Other: LifeScience Technologies application

INTERVENTIONS:
Other: LifeScience Technologies application — Application for mobile devices. The app enables users to review educational videos about a surgery and recovery from a surgery from home. It also enables the user to track different metrics specific to the user's health.
  Other Names: LST app

SUMMARY:
The purpose of this study is to learn whether it is feasible to use the LifeScience Technologies application (LST app) in patients undergoing radical cystectomy with the eventual goal to reduce complications and readmissions to the hospital after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent Non-muscle invasive bladder cancer (NMIBC) or Muscle-invasive Bladder Cancer (MIBC) and are candidates for radical cystectomy
* Subjects must have an internet connection and be able and willing to use an applicable device. If patients do not have an applicable device, they must be willing to borrow an iPad from the study team (to be returned at the conclusion of the study).

Exclusion Criteria:

* No internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2018-02-14 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Compliance using LST app at home | 90 Days
  The LST app logs user activity. The study team will track user compliance with completing forms and questions within the application.

SECONDARY OUTCOMES:
Patient-generated subjective global assessment (PG-SGA) | Baseline
  Test the PG-SGA using the LST app to see if it is feasible in practice at identifying patients at increased risk of malnutrition.
Edmonton Frail Scale (EFS) | Baseline
  Test the EFS using the LST app to see if it is feasible in practice at identifying frail patients.
Physician Office/Clinician and Group Consumer Assessment of Healthcare Providers and Systems (CG-CAHPS) Survey Research (HealthStream™) | Change from Baseline to Day 90
  Measure of how well the patient understood the various tests and procedures that were discussed with them before and after surgery.
Count of readmissions | Day 90
  Count of the number of readmissions to the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Lee, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States